CLINICAL TRIAL: NCT01806220
Title: Laryngeal and Esophageal EGF-r Expression in Patients With Reflux Laryngitis
Acronym: EGFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, CLAUDIA ALESSANDRA ECKLEY, Professor Otolaryngology Department, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: fcmscsp180/06
Record Dates: First submitted 2012-08-29; First posted 2013-03-07 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Gastroesophageal Reflux Disease; Chronic Laryngitis
Keywords: Gastroesophageal Reflux Disease (GERD); Chronic Laryngitis; Epidermal Growth factor receptor
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- biopsy of retrocrycoid laryngeal mucosa (Active Comparator): During upper digestive endoscopy a biopsy specimen of the retrocrycoid laryngeal mucosa was obtained with a forceps introduced by the working channel of the scope.
  Intervention: biopsy of retrocrycoid laryngeal mucosa
  Interventions: Procedure: Biopsy of the retrocrycoid laryngeal mucosa
- biopsy of distal esophagus mucosa (Active Comparator): during upper digestive endoscopy a biopsy specimen of the distal esophageal mucosa was obtained
  Intervention:biopsy of distal esophagus mucosa
  Interventions: Procedure: Biopsy of the distal esophageal mucosa

INTERVENTIONS:
Procedure: Biopsy of the retrocrycoid laryngeal mucosa — Biopsies of the retrocrycoid laryngeal mucosa were performeed under sedation using a forceps introduced by the working channel of the endoscope
  Arms: biopsy of retrocrycoid laryngeal mucosa
Procedure: Biopsy of the distal esophageal mucosa — Biopsies were performeed under sedation using a forceps introduced by the working channel of the endoscope during upper digestive endoscopy
  Arms: biopsy of distal esophagus mucosa

SUMMARY:
* Saliva plays an important role in the homeostasis of the digestive tract mucosa.
* Salivary organic components, such as the Epidermal Growth Factor(EGF) have been found in defficient concentrations in patients with gastroesophageal reflux disease (GERD) and reflux related laryngitis (LPR).
* The epidermal growth factor receptor (EGFR) signaling pathway is one of the most important pathways that regulate growth, survival, proliferation, and differentiation in mammalian cells
* Eperdermal growth factor receptor (EGFR) overexpression has been linked to hyperproliferative diseases.
* It is unknown if the inflammatory process in GERD is realated to difficiencies in EGFR expression.
* The objective of the current study was to try to establish a correlation between the expression of EGFR in the laryngeal and esophageal mucosa and the severity of laryngitis in adults with GERD and LPR

DETAILED DESCRIPTION:
Objectives: The expression of the Epidermal Growth Factor receptor (EGFR) has been studied in a number of neoplastic and chronic diseases, but there are no reports in literature regarding its expression in chronic laryngitis associated to Gastroesophageal Reflux isease (GERD), also known as Laryngopharyngeal Reflux (LPR). The current study compared the expression of EGFR in the esophageal and laryngeal mucosa of adults with GERD and LPR. Study Design: Prospective based on imunohistochemical analysis of parafine embedded biopsy specimens and clinical data. Methods: From August, 2004 to February 2007 a total of 24 adults with confirmed diagnosis of LPR and no other clinical conditions or habits known to cause chronic laryngitis were studied at a University Hospital. Biopsies of the distal esophagus and the retrocrycoid laryngeal mucosa were obtained during upper digestive endoscopy. Data were analyzed statistically comparing samples in each individual and between individuals using the severity of histological signs of inflammation on hematoxacillin and eosinophillin (HE) stains to immunohistochemical analysis of the expression of EGFR. Other independent variables were severity of symptoms and signs, gender and age. Fishers´s exact test and multivariance ANOVA tests were used with significance level established at 95%.

ELIGIBILITY:
Inclusion Criteria:

* Adults with reflux laryngitis diagnosed by clinical symptoms (Reflux Symptom -Index >13) and videolaryngoscopic signs (Reflux Finding Score >7)
* A positive 24-hour doube probe esophageal ph monitoring test

Exclusion Criteria:

* Other known causes of chronic laryngitis or inflammatory conditions of the pharynx, larynx and upper digestive tract.
* Current or past history of Head and Neck or digestive tract tumors.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Epidermal Growth Factor Receptor (EGFR) expression in laryngeal and esophageal mucosa of patients with chronic reflux laryngitis | prospective study that enrolled every adult patient with reflux laryngitis and no other causes of chronic laryngeal and pharyngeal inflammation during a 36 month period
  Patients with reflux laryngitis diagnosed by suggestive symptoms (Reflux Symptom Index>13) and videolaryngoscopic signs (Reflux Finding Score>7) and confirmed by a 24-hour double probe esophageal ph monitoring test were consecutively enrolled properly informed and consented.

SECONDARY OUTCOMES:
Compare Epidermal Growth Factor Receptor expression in different severities of inflammatory responses. | EGFR expression of the esophageal and laryngeal mucosas was compared to clinical, videolaryngoscopic and microscopic inflammatory signs. (up to 36 months)
  Mucosal biopsy specimens obtained during routine upper digestive tract endocopic examination under sedation were obtained.

CONTACTS AND LOCATIONS:
Overall Officials: CLAUDIA A ECKLEY, MD, Principal Investigator — SANTA CASA SCHOOL OF MEDICINE AND HOSPITALS OF SÃO PAULO BRAZIL
Locations (1):
- Santa Casa School of Medicine and Hospitals of São Paulo Brazil, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Eckley CA, Michelsohn N, Rizzo LV, Tadokoro CE, Costa HO. Salivary epidermal growth factor concentration in adults with reflux laryngitis. Otolaryngol Head Neck Surg. 2004 Oct;131(4):401-6. doi: 10.1016/j.otohns.2004.01.020. PMID 15467608
- [Background] Eckley CA, Rios Lda S, Rizzo LV. Salivary egf concentration in adults with reflux chronic laryngitis before and after treatment: preliminary results. Braz J Otorhinolaryngol. 2007 Mar-Apr;73(2):156-60. doi: 10.1016/s1808-8694(15)31060-0. PMID 17589721
- [Background] Sarosiek J, McCallum RW. Do salivary organic components play a protective role in health and disease of the esophageal mucosa? Digestion. 1995;56 Suppl 1:32-7. doi: 10.1159/000201299. PMID 7556968
- [Background] Rourk RM, Namiot Z, Edmunds MC, Sarosiek J, Yu Z, McCallum RW. Diminished luminal release of esophageal epidermal growth factor in patients with reflux esophagitis. Am J Gastroenterol. 1994 Aug;89(8):1177-84. PMID 8053431